CLINICAL TRIAL: NCT02199808
Title: Fatty Acids and Executive Functions: Cortical Activation and Behavioral Performance.
Brief Title: Fatty Acids and Executive Function Development in 7-12 Year Olds
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Sigma Xi (Unknown)
Responsible Party: Principal Investigator, Carol Cheatham, PhD, Associate Professor of Psychology & Neuroscience, University of North Carolina, Chapel Hill
Other Study IDs: 14-0198
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Executive Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 7-9 year olds: These are children who are between 7 and 9 years old when they are tested.
- 10-12 year olds: These are children who are between 10 and 12 years old when they are tested.

SUMMARY:
Purpose: To examine the effect of the omega-6 to omega-3 fatty acid ratio on age-related changes in executive functions in children and older adults.

Participants: Eighty-four typically-developing 7-to 12-year-old children.

Procedure (methods): Participants and a caregiver will participate in 4 sessions. Three sessions will consist of the screening. These sessions will be telephone calls to collect 24-hour diet information that will be used to determine whether they are eligible for the fourth session. Approximately 120 participants will be screened to find 84 participants who are eligible for the fourth session, in which participants will complete a series of tests on the Cambridge Neuropsychological Test Automated Battery (CANTAB) - a touch-screen device that provides computerized versions of standardized cognitive tests. They will also complete a maze task in which they figure out a path through the maze by walking on the correct squares. Brain activity will be recorded using a portable near-infrared spectroscopy (NIRS) system.

ELIGIBILITY:
Inclusion Criteria:

* Typically-developing children 7-12 years old

Exclusion Criteria:

* Children or parents who do not speak English
* Any diagnosis of a psychological illness
* History of seizures
* History of tobacco exposure during gestation
* History of alcohol exposure during gestation

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All participants will be typically-developing, healthy 7-to-12-year-olds who are fluent in English. Every effort will be made to recruit roughly equal numbers of boys and girls. Recruitment will be conducted irrespective of race and ethnicity. An attempt will be made to match the sample to the race and ethnicity of the region: 80% White, 15% African-American, and 5% Native American, Asian, and Other descent.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Error (count) and latency (in milliseconds) measures from executive function tasks | One time with children who are 7-12 years old
  For one specific aim, the omega-6 to omega-3 fatty acid ratio will be determined by summing the omega-6 and omega-3 fatty acid levels in plasma and dividing omega-6 fatty acids by omega-3 fatty acids. The calculated ratio will be used to predict error and latency scores on executive function tasks.
  For a second specific aim, the oxygenated and deoxygenated hemoglobin concentrations from near-infrared spectroscopy (NIRS) measurements will be used to predict the error and latency measures from executive function tasks.

SECONDARY OUTCOMES:
Oxygenated and deoxygenated hemoglobin concentrations from near-infrared spectroscopy (NIRS) | One time with children who are 7-12 years old.
  Plasma levels of omega-6 and omega-3 fatty acids will be used to predict oxygenated and deoxygenated hemoglobin concentrations from near-infrared spectroscopy (NIRS) measurements in children who are 7-12 years old.
Performance on the Maze as measured by Noldus Ethovision | One time with children who are 7-12 years old
  Performance on the Maze as measured by Noldus Ethovision tracking system will be compared to performance on standardized measures of planning and spatial working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill's Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Ingol TT, Li R, Boone KM, Rausch J, Klebanoff MA, Turner AN, Yeates KO, Nelin MA, Sheppard KW, Keim SA. Docosahexaenoic and Arachidonic Acid Supplementation of Toddlers Born Preterm Does Not Affect Short-Term Growth or Adiposity. J Nutr. 2019 Dec 1;149(12):2182-2190. doi: 10.1093/jn/nxz115. PMID 31187863
- [Derived] Sheppard KW, Cheatham CL. Omega-6/omega-3 fatty acid intake of children and older adults in the U.S.: dietary intake in comparison to current dietary recommendations and the Healthy Eating Index. Lipids Health Dis. 2018 Mar 9;17(1):43. doi: 10.1186/s12944-018-0693-9. PMID 29523147
- [Derived] Sheppard KW, Cheatham CL. Executive functions and the omega-6-to-omega-3 fatty acid ratio: a cross-sectional study. Am J Clin Nutr. 2017 Jan;105(1):32-41. doi: 10.3945/ajcn.116.141390. Epub 2016 Nov 16. PMID 27852615